CLINICAL TRIAL: NCT01585207
Title: Open Label Safety and Tolerability Trial of CPP-109 (Vigabatrin) in Adults With Treatment Refractory Tourette's Disorder
Brief Title: Proof-of-Concept Safety Study of CPP-109 (Vigabatrin) for Treatment Refractory Tourette's Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barbara J. Coffey (Other)
Responsible Party: Sponsor-Investigator, Barbara J. Coffey, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-0964; 11-01864
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Tourette's Disorder
Keywords: Tourette's Disorder; vigabatrin
MeSH Terms: conditions — Tourette Syndrome | interventions — Vigabatrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vigabatrin (Experimental): 3 tablets, bid for 8 weeks
  Interventions: Drug: vigabatrin

INTERVENTIONS:
Drug: vigabatrin — 3 tablets, bid for 8 weeks
  Other Names: CPP-109 Vigabatrin

SUMMARY:
The purpose of this study is to determine if vigabatrin, an unusual anti-seizure medication, will diminish the Tourette Disorder outbursts in young adults whose symptoms have persisted into adulthood and have not responded to usual treatment.

DETAILED DESCRIPTION:
The aims of this study are to 1) explore proof of concept that CPP-109 will reduce tics, and 2) to obtain systematic data regarding dosing, safety and tolerability of CPP-109 in adults with treatment refractory TD. We will obtain preliminary data on estimate of effect size for tics using Cohen's d, calculating the difference between the two means (baseline and endpoint scores on the YGTSS), divided by the standard deviation of the difference.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 and 35 years of age (inclusive) when informed consent is obtained.
2. Subjects must meet full DSM-IV diagnostic criteria for TD by clinical interview on examination by a physician investigator, and confirmed by the Structured Clinical Interview for DSM (SCID-CT) for clinical trials.
3. Subjects will have failed to respond to an adequate trial, as determined by the investigator, of clonidine, guanfacine, and a first generation (typical) and second-generation (atypical) neuroleptic medication in the past.
4. Tics are causing significant distress or impairment, as determined by the subject and principal investigator, on the current treatment regimen.
5. Laboratory results, including serum chemistries, hematology, and urinalysis, must show no significant abnormalities (significant is defined as laboratory values requiring acute medical intervention).
6. Subjects will not undergo formal IQ testing, but must be of normal intelligence in the judgment of the investigator.
7. Subjects must possess an educational level, degree of understanding and command of the English language to enable them to communicate suitably with the investigators and study coordinator, and to understand the nature of the study.
8. Subjects must be considered reliable.
9. Written informed consent of subjects is obtained.

Exclusion Criteria:

1. Subjects with organic brain disease, for example, traumatic brain injury residua.
2. Subjects with a preexisting ophthalmologic condition.
3. Subjects with or at high risk of other types of irreversible vision loss or who require other drugs associated with serious adverse ophthalmic effects such as retinopathy or glaucoma.
4. Subjects meeting criteria for mental retardation as defined by the DSM-IV-TR.
5. Subjects with a history of seizure disorder (other than febrile seizure).
6. Subjects with history of Sydenham's Chorea.
7. Subjects with autism, schizophrenia, other psychotic disorder, or bipolar disorder.
8. Subjects with a primary diagnosis of a major mood disorder that requires ongoing psychiatric treatment.
9. Subjects with a neurological disorder other than a tic disorder.
10. Subjects with a major medical illness.
11. Female subjects who are unwilling to use birth control or who are pregnant, as determined by serum pregnancy test at baseline assessment, or lactating.
12. Subjects who have a past or current history of substance dependence and/or a current history of substance abuse or who fail baseline toxicology screen.
13. Subjects who have any clinically significant abnormal laboratory result at baseline screening including EKG, or blood tests.
14. Subjects who, in the opinion of the investigator, are unsuitable in any other way to participate in this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Brodie, PhD,MD, Principal Investigator — NYU School of Medicine
Locations (1):
- Tics and Tourette's Clinical and Research Program, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vigabatrin
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vigabatrin
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 34.75 [26 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
YGTSS (total tic) [Mean (Standard Deviation); unit: total tics] — Yale Global Tic Severity Scale (YGTSS) - The Total Tic Score is a summation of the Total Motor Tic (0 -25) and Total Phonic Tic (0-25) Scores, full range 0 (No impairment) to 50 (Severe impairment)
  total tics | 39 (3.67)

OUTCOME MEASURES:

1. Primary Outcome: Global Severity Score on the Y-GTSS
Description: The Global Severity score is the sum of the Total Tic score and the TD Impairment score. It is rated by the Investigator on the Yale Global Tic Severity Score ( Y-GTSS, a widely accepted measure of drug efficacy in TD. Scale from 0- 100. Higher score indicates more impairment.
Time Frame: weekly from baseline to end of study (10weeks)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vigabatrin
Number analyzed (Participants) | 4
units on a scale
  Baseline | 80.25 [76 to 90]
  Week 0 | 78.75 [75 to 83]
  Week 1 | 61 [36 to 77]
  Week 2 | 69.75 [63 to 78]
  Week 3 | 61 [57 to 68]
  Week 4 | 59 [49 to 65]
  Week 6 | 58.75 [44 to 68]
  Week 8 | 60.88 [44 to 69.5]
  Week 10 | 70.33 [53 to 86]

ADVERSE EVENTS:
Arm/Group | Vigabatrin
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vigabatrin (N=4)
Fatigue (General disorders) | 3
Appetite Increase (General disorders) | 1
Sleep Difficulties (General disorders) | 1
Increase in OCD symptoms (Nervous system disorders) | 1
Dry mouth (General disorders) | 1
Mood swings (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Daytime tiredness (General disorders) | 1
Vivid dreams (General disorders) | 1
Possible weight gain (General disorders) | 1
Blurry Vision (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No